CLINICAL TRIAL: NCT06138613
Title: Motion Delos: An Open Label Study to Investigate the Safety and Efficacy of Tradipitant in Participants Affected by Motion Sickness During Travel
Brief Title: Motion Delos: An Open Label Safety and Efficacy of Tradipitant in Participants Affected by Motion Sickness
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-VLY-686-3403
Record Dates: First submitted 2023-03-03; First posted 2023-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant Dose A (Experimental): "See Drug"
  Interventions: Drug: Tradipitant
- Tradipitant Dose B (Experimental): "See Drug"
  Interventions: Drug: Tradipitant

INTERVENTIONS:
Drug: Tradipitant — Oral Capsule

SUMMARY:
An open label study to investigate the safety and efficacy of tradipitant in participants affected by motion sickness during travel

DETAILED DESCRIPTION:
This is an open label study to investigate the efficacy and safety of tradipitant in motion sickness affected male and female participants during events historically known to cause motion sickness.

ELIGIBILITY:
Inclusion Criteria:

* History of Motion Sickness
* Age 18-75

Exclusion Criteria:

* Nausea-inducing disorder other than motion sickness
* BMI > 40
* History of intolerance and/or hypersensitivity to Neurokinin-1 Receptor antagonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of tradipitant as measured by reporting of adverse events (AEs). | through study completion, approximately 1 year
  Safety will be monitored using clinical measures, vital signs, blood chemistry, hematology, urology, and ECGs.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Monica Clinical Trials, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No